CLINICAL TRIAL: NCT01820936
Title: Open-Label, Randomized, 4-Way Crossover Study to Determine the Effect of Food on the Pharmacokinetics of PCI-32765
Brief Title: A Study to Determine the Effect of Food on the Pharmacokinetics of PCI-32765
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR101204; PCI-32765CLL1001 (Other: Janssen Research & Development, LLC); 2013-000963-96 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-29 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; PCI-32765; PCI-45227; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A: PCI-32765 (Experimental): 420 mg capsules administered by mouth with 240 mL noncarbonated water 30 minutes after completing a high-fat breakfast
  Interventions: Drug: Sequence 1: PCI-32765; Drug: Sequence 2: PCI-32765; Drug: Sequence 3: PCI-32765; Drug: Sequence 4: PCI-32765
- Treatment B: PCI-32765 (Experimental): 420 mg capsules administered by mouth with 240 mL noncarbonated water after fasting for at least 10 hours and 30 minutes before starting a high-fat breakfast
  Interventions: Drug: Sequence 1: PCI-32765; Drug: Sequence 2: PCI-32765; Drug: Sequence 3: PCI-32765; Drug: Sequence 4: PCI-32765
- Treatment C: PCI-32765 (Experimental): 420 mg capsules administered by mouth with 240 mL noncarbonated water 2 hours after completing a high-fat breakfast
  Interventions: Drug: Sequence 1: PCI-32765; Drug: Sequence 2: PCI-32765; Drug: Sequence 3: PCI-32765; Drug: Sequence 4: PCI-32765
- Treatment D: PCI-32765 (Experimental): 420 mg capsules administered with 240 mL noncarbonated water after fasting at least 10 hours
  Interventions: Drug: Sequence 1: PCI-32765; Drug: Sequence 2: PCI-32765; Drug: Sequence 3: PCI-32765; Drug: Sequence 4: PCI-32765
- Treatment E: PCI-32765 (Experimental): 840 mg capsules administered with 240mL noncarbonated water 30 minutes after completing a high-fat breakfast
  Interventions: Drug: Sequence 5: PCI-32765

INTERVENTIONS:
Drug: Sequence 1: PCI-32765 — Period 1 = Treatment D, Period 2 = Treatment C, Period 3 = Treatment A, Period 4 = Treatment B
  Arms: Treatment A: PCI-32765; Treatment B: PCI-32765; Treatment C: PCI-32765; Treatment D: PCI-32765
Drug: Sequence 2: PCI-32765 — Period 1 = Treatment A, Period 2 = Treatment D, Period 3 = Treatment B, Period 4 = Treatment C
  Arms: Treatment A: PCI-32765; Treatment B: PCI-32765; Treatment C: PCI-32765; Treatment D: PCI-32765
Drug: Sequence 3: PCI-32765 — Period 1 = Treatment B, Period 2 = Treatment A, Period 3 = Treatment C, Period 4 = Treatment D
  Arms: Treatment A: PCI-32765; Treatment B: PCI-32765; Treatment C: PCI-32765; Treatment D: PCI-32765
Drug: Sequence 4: PCI-32765 — Period 1 = Treatment C, Period 2 = Treatment B, Period 3 = Treatment D, Period 4 = Treatment A
  Arms: Treatment A: PCI-32765; Treatment B: PCI-32765; Treatment C: PCI-32765; Treatment D: PCI-32765
Drug: Sequence 5: PCI-32765 — After completion of the 4-way crossover, an additional separate cohort of 8 subjects were enrolled. These subjects participated in 1 treatment period to document safety and PK
  Arms: Treatment E: PCI-32765

SUMMARY:
The purpose of this study is to compare the effect of food and two modified fasting regimens on the pharmacokinetics (study of what the body does to a drug) of PCI-32765 in healthy adult participants.

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned by chance to study treatments), open-label (identity of assigned study drug will be known), 4-way crossover study to compare the effect of food and two fasting regimens on the pharmacokinetics of PCI-32765 in healthy adults. There will be approximately 52 (at least 25% women) participants (11 in each sequence in the 4-way crossover and 8 in an optional cohort). A screening phase will be followed by an open-label treatment phase consisting of 4 single-dose treatment periods of 420 mg PCI-32765 administered with or without food. Doses in successive open-label treatment periods will be separated by a washout period of 7 days. Participants will be confined to the study center from Day -1 of each treatment period (at least 10 hours before each study drug administration) until completion of the 72 hour pharmacokinetic blood sample collection on Day 4 of Period 4. Blood samples for pharmacokinetic analysis of PCI-32765 and metabolite PCI-45227 will be collected before dosing and over 72 hours after dosing in each treatment period. A follow-up visit approximately 10 days after the last dose will be made to measure lymphocyte count and to capture any additional adverse events. After completion of the 4-way crossover portion of the study, and in absence of significant safety observations at the 420 mg PCI-32765 dose, an additional separate cohort of 8 participants may be enrolled to participate in one treatment period and receive a dose of 840 mg in combination with a high-fat breakfast. Safety will be assessed throughout the study. The total study duration is a maximum of 85 days.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal or documented as surgically sterile
* Men must agree to use an adequate contraception method as deemed appropriate by the investigator during the study and for 3 months after receiving the last dose of study drug, and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index between 18 and 30 kg/m2and body weight not less than 50 kg
* Blood pressure (after sitting for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, history of immune disorders (eg, lupus, rheumatoid arthritis, psoriatic arthritis) or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, PFA-100, clinical chemistry or urinalysis at screening
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening
* Use of aspirin, non-steroidal anti-inflammatory agents, clopidogrel, Vitamin E supplements, fish oil, or flax seed within 1 week before PFA-100 assay test at screening
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, and hormonal replacement therapy, within 14 days before the first dose of the study drug is scheduled
* Use of herbal supplements (such as St. John's Wort) within 30 days of the first dose administration
* Has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 2 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines) at screening and Day -1 of each treatment period
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics
* Known allergy to the study drug or any of the excipients of the formulation
* Known allergy to heparin or history of heparin induced thrombocytopenia
* Donated blood or blood products or had substantial loss of blood within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies
* History of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or participant's verbal report and confirmed by cotinine test
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentrations of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Area under the plasma concentration-time curve from time 0 to infinite time of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Maximum plasma concentration of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours

SECONDARY OUTCOMES:
Time to reach the maximum plasma concentration of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Elimination half-life of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Relative bioavailability of PCI-32765 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
  Relative bioavailability is defined as the ratio of the area under the concentration curve to infinity between the test treatment and the reference treatment.
Maximum plasma concentration of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Time to reach the maximum plasma concentration of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentrations of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Area under the plasma concentration-time curve from time 0 to infinite time of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Elimination half-life of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Relative bioavailability of metabolite PCI-45227 | Predose; postdose at 30 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours
Number of participants with adverse events | Up to 30 days following the last dose of study drug
Number of participants with adverse events of special interest (major hemorrhage and intracranial hemorrhage) | Up to 30 days following the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States

REFERENCES:
- [Derived] de Jong J, Sukbuntherng J, Skee D, Murphy J, O'Brien S, Byrd JC, James D, Hellemans P, Loury DJ, Jiao J, Chauhan V, Mannaert E. The effect of food on the pharmacokinetics of oral ibrutinib in healthy participants and patients with chronic lymphocytic leukemia. Cancer Chemother Pharmacol. 2015 May;75(5):907-16. doi: 10.1007/s00280-015-2708-9. Epub 2015 Feb 28. PMID 25724156
- See also: Open-Label, Randomized, 4-Way Crossover Study to Determine the Effect of Food on the Pharmacokinetics of PCI-32765 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3872&filename=CR101204_CSR.pdf